CLINICAL TRIAL: NCT02279251
Title: School Based Low-intensity Cognitive Behavioral Intervention for Anxious Youth. A Randomized Controlled Trial
Brief Title: School Based Low-intensity Cognitive Behavioral Intervention for Anxious Youth
Acronym: LIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: The Research Council of Norway (Other); Modum Bad (Other); Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 229020
Record Dates: First submitted 2014-10-15; First posted 2014-10-31 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Anxiety
Keywords: Anxiety; adolescents; school-based; low-intensity CBT
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief CBT (VÅG) (Active Comparator): This is a brief five session CBT group intervention developed at Uni Research. The intervention include self-help material (Psychological First Aid) for the adolescents to use at home between sessions.
  Interventions: Behavioral: VÅG
- Established CBT program (Cool Kids) (Active Comparator): An established, 10 session CBT group program (school version) developed by researchers at Macquarie University, Australia. The intervention has previously not been evaluated with Norwegian adolescents.
  Interventions: Behavioral: CHILLED
- Waitlist (No Intervention): Waiting period is ten weeks, then participants are randomized to one of the two active interventions

INTERVENTIONS:
Behavioral: VÅG — Low-intensity CBT intervention
  Arms: Brief CBT (VÅG)
Behavioral: CHILLED — Standard length CBT intervention
  Arms: Established CBT program (Cool Kids)

SUMMARY:
The study will evaluate two group CBT interventions delivered by school health nurses, in cooperation with community psychologist and mental health care personnel, to adolescents with mild to moderate levels of anxiety symptoms. The two interventions have different intensity (5 versus 10 group meetings). The two group interventions will be compared to a waitlist control group.

DETAILED DESCRIPTION:
Anxiety disorders are among the major mental health problems in children and adolescents, with regard to prevalence and long-term consequences. Cognitive behavioural therapy (CBT) has proven to be effective as treatment, early intervention and prevention of youth anxiety disorders. The majority of youth with anxiety problems, however, is not in contact with mental health services and do not receive effective help. This is due to shortage of personnel, resources and time among mental health-personal delivering treatment, as well as health services not being easily accessable for adolescents. School-based, low-intensity early intervention programs (indicated prevention) may improve access to effective treatment for youth with internalizing problems, and also promote more effective use of health services. The present study is a multi-site randomized controlled study with early intervention to be conducted within the primary health care service in three parts of Norway; including nine municipalities from west, east and south of Norway. A brief CBT program will be compared to a longer CBT program, and a wait-list control group. The effects will be evaluated with regard to decrease in youth internalizing symptoms. The CBT interventions are given to adolescents with mild to moderate levels of anxiety symptoms. Interventions are delivered by trained school-health nurses in collaboration with and/or supervised by experienced CBT therapists. The study involves researchers from three research environments in Norway, and collaboration with prominent international researchers from USA and Australia.The study has potential impact on how to deliver effective low-threshold interventions to anxious youth.

ELIGIBILITY:
Inclusion Criteria:

1. An overall score of > 25 on the anxiety inventory Spence Children's Anxiety Scale (SCAS) and a score of > 1 on the first question of the Children's Anxiety Life Interference Scale (CALIS), indicating that anxiety interferes with daily life of the youth, rated either by the adolescents or by one parent.
2. The adolescent and at least one parent understand and read Norwegian.
3. Assent from the youth and signed informed consent from the parent.

Exclusion Criteria:

The adolescent has a behavior that makes participation in groups with other adolescents challenging. This is evaluated by the school nurse, based on information from the adolescent, the parent and the teacher. In each case, the school nurse makes an evaluation based on the following questions:

1. Is the adolescent able to follow group-rules?
2. Will the adolescent behave in ways that disrupts the group?
3. Does the adolescent have learning problems to an extent that will make it difficult to follow the group program?

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 313 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Spence Children's Anxiety Scale | Changes from baseline to 4 weeks, 10 weeks, and 1 year
  Self-reported (child and parent version) child anxiety symptoms, 38 items questionnaire, rated at a 4-point scale.
Children Anxiety Life Interference Scale | Changes from baseline to 4 weeks,10 weeks, and 1 year
  Self-reported (child and parent version) of degree of life interference of child anxiety symptoms

SECONDARY OUTCOMES:
Short Mood and Feeling Questionnaire | Changes from baseline to 4 weeks,10 weeks,and 1 year
  Questionnaire measuring symptoms of depression (child and parent version)
Questionnaire for Measuring Health-Related Quality of Life Children and Adolescents (KINDL-R) | Changes from baseline to 10 weeks, and 1 year
  Questionnaire (child and parents version) measuring quality of life in youth
Clinical Global Impression Scale, severity/improvement (CGI-S/I) | Changes from baseline to 10 weeks, and 1 year
  The clinician's (i.e. the school health nurse) global assessment of level of youth anxiety
Sleep problems | Changes from baseline, up to 10 weeks, and after 1 year
  Questionnaire (youth) on variables related to sleep (sleep duration, insomnia etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Bente Storm Mowatt Haugland, PhD, Principal Investigator — Uni Research Health
Locations (3):
- Norway (3):
  - Municipality of Modum, Oslo, East Norway
  - Municipality of Fjell, Sund and Askoy, Fjell
  - Sorlandet Hospital HF, Kristiansand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haugland BSM, Haaland AT, Baste V, Bjaastad JF, Hoffart A, Rapee RM, Raknes S, Himle JA, Husabo E, Wergeland GJ. Effectiveness of Brief and Standard School-Based Cognitive-Behavioral Interventions for Adolescents With Anxiety: A Randomized Noninferiority Study. J Am Acad Child Adolesc Psychiatry. 2020 Apr;59(4):552-564.e2. doi: 10.1016/j.jaac.2019.12.003. Epub 2020 Jan 8. PMID 31926224
- [Result] Haugland BS, Raknes S, Haaland AT, Wergeland GJ, Bjaastad JF, Baste V, Himle J, Rapee R, Hoffart A. School-based cognitive behavioral interventions for anxious youth: study protocol for a randomized controlled trial. Trials. 2017 Mar 4;18(1):100. doi: 10.1186/s13063-017-1831-9. PMID 28259171
- [Result] Haugland BSM, Hysing M, Baste V, Wergeland GJ, Rapee RM, Hoffart A, Haaland AT, Bjaastad JF. Sleep Duration and Insomnia in Adolescents Seeking Treatment for Anxiety in Primary Health Care. Front Psychol. 2021 Mar 24;12:638879. doi: 10.3389/fpsyg.2021.638879. eCollection 2021. PMID 33841272
- [Result] Haugland BSM, Hysing M, Hoffart A, Haaland AT, Bjaastad JF, Wergeland GJ, Baste V. Effect of early intervention for anxiety on sleep outcomes in adolescents: a randomized trial. Eur Child Adolesc Psychiatry. 2022 Oct;31(10):1-15. doi: 10.1007/s00787-021-01795-6. Epub 2021 May 7. PMID 33961115